CLINICAL TRIAL: NCT05630027
Title: Soothing and Anti-hair Loss Activity of a Scalp Lotion Containing Piroctone Olamine, 2,4 Diaminopyrimidine Oxide and Vichy Mineralizing Water
Brief Title: A Scalp Lotion Toimprove Sensitive Scalp Syndrome
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: AC5+
Record Dates: First submitted 2022-11-18; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Alopecia; Sensitive Skin
Keywords: alopecia; sensitive skin; prurit
MeSH Terms: conditions — Alopecia | interventions — piroctone olamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Piroctone Olamine (PO), 2,4 Diaminopyrimidine oxide (2.4 DA) and Vichy mineralizing water — observational, prospective study

SUMMARY:
Overall, 100 Caucasian subjects participated in this 6-weeks lasting study, AC5+ was applied daily. All subjects had clinically confirmed mild to moderate alopecia and self-declared sensitive scalp. Instrumental assessments included Trans Epidermal Water Loss (TEWL), inflammation markers, clinical assessments included the severity of erythema, inflammation and greasiness. Subjective/Self assessments comprised the intensity of the scalp itch/pruritus and the evaluation of their head hair status (volume, abundance, strength). Same assessments were provided by the investigators.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* mild alopecia:
* female: Ludwig type 1
* male: Hamilton III to IV type

Exclusion Criteria:

* Moderate or severe alopecia
* Dandruff

Age Groups: Child, Adult, Older Adult
Study Population: Adult subjects with mild alopecia and no dandruff
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
erythema | Baseline
  on a scale from o=none to 5=severe
erythema | Day 21
  on a scale from o=none to 5=severe
inflammation | Baseline
  on a scale from o=none to 5=severe
inflammation | Day 21
  on a scale from o=none to 5=severe
greasiness | Baseline
  on a scale from o=none to 5=severe
greasiness | Day 21
  on a scale from o=none to 5=severe
Global soothing score | Baseline
  sum of the symptoms with a score up to 15
Global soothing score | Day 21
  sum of the symptoms with a score up to 15

SECONDARY OUTCOMES:
pruritus | Baseline
  on a scale from o=none to 5=severe
pruritus | Day 21
  on a scale from o=none to 5=severe
burning | Baseline
  on a scale from o=none to 5=severe
burning | Day 21
  on a scale from o=none to 5=severe
stinging | Baseline
  on a scale from o=none to 5=severe
stinging | Day 21
  on a scale from o=none to 5=severe
scratching | Baseline
  on a scale from o=none to 5=severe
scratching | Day 21
  on a scale from o=none to 5=severe
hair quality | Baseline
  on a scale from o=none to 5=severe
hair quality | Day 21
  on a scale from o=none to 5=severe
Transepidermal water loss | Baseline
  instrumental measurements
Transepidermal water loss | Day 21
  instrumental measurements
Inflammation markers | Baseline
  skin swabs analysis
Inflammation markers | Day 21
  skin swabs analysis skin swabs analysis
squalene | Baseline
  skin swabs analysis skin swabs analysis
squalene | Day 21
  skin swabs analysis skin swabs analysis
Squalene monohydroperoxide | Baseline
  skin swabs analysis
Squalene monohydroperoxide | Day 21
  skin swabs analysis

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Massiot, Study Director — L'OREAL Research and Innovation, Saint-Ouen, France
Locations (1):
- L'OREAL Research and Innovation, Saint-Ouen, France

IPD SHARING:
Plan to Share IPD: No